CLINICAL TRIAL: NCT05058066
Title: Long-term Follow-up of a Wide Diameter Bone Anchored Hearing Implant: the 10-year Experience on Stability, Survival and Tolerability of the BIA300®
Brief Title: 10-year Follow-up of a Wide Diameter Bone Anchored Hearing Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAG5173/CBAS5562 10y
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2021-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control implant loaded at 6 weeks post-surgery (Active Comparator): The control implant included the previous generation as-machined titanium Baha® flange fixture (diameter 3.75mm; length 4mm) with 6mm conically shaped abutment.
  Interventions: Device: Baha® flange fixture (diameter 3.75mm; length 4mm) with 6mm abutment
- Test implant loaded at 6 weeks post-surgery (Experimental): The test implant and the implant used for the 3-week loading trial included the wide diameter titanium implant (diameter 4.5mm; length 4mm) with 6mm rounded, apically converging titanium abutment developed by Cochlear Bone Anchored Solutions AB (Mölnlyncke, Sweden). This system with an additional minor change to the internal abutment connection design was later commercialized under the name Cochlear™ Baha® BIA300 Implant with abutment.
  Interventions: Device: Baha® BIA300 Implant (diameter 4.5mm; length 4mm) with 6mm abutment
- Test implant loaded at 3 weeks post-surgery (Experimental): The test implant and the implant used for the 3-week loading trial included the wide diameter titanium implant (diameter 4.5mm; length 4mm) with 6mm rounded, apically converging titanium abutment developed by Cochlear Bone Anchored Solutions AB (Mölnlyncke, Sweden). This system with an additional minor change to the internal abutment connection design was later commercialized under the name Cochlear™ Baha® BIA300 Implant with abutment.
  Interventions: Device: Baha® BIA300 Implant (diameter 4.5mm; length 4mm) with 6mm abutment; Procedure: Early loading

INTERVENTIONS:
Device: Baha® flange fixture (diameter 3.75mm; length 4mm) with 6mm abutment — The control implant included the previous generation as-machined titanium Baha® flange fixture (diameter 3.75mm; length 4mm) with 6mm conically shaped abutment.
  Arms: Control implant loaded at 6 weeks post-surgery
Device: Baha® BIA300 Implant (diameter 4.5mm; length 4mm) with 6mm abutment — The test implant and the implant used for the 3-week loading trial included the wide diameter titanium implant (diameter 4.5mm; length 4mm) with 6mm rounded, apically converging titanium abutment developed by Cochlear Bone Anchored Solutions AB (Mölnlyncke, Sweden). This system with an additional minor change to the internal abutment connection design was later commercialized under the name Cochlear™ Baha® BIA300 Implant with abutment. In addition to the difference in abutment shape and the wider diameter, the test implant incorporates small-sized threads at the implant neck and the moderately rough TiOblast™ (Dentsply, Mölndal, Sweden) surface on the intraosseous part of the implant6-8.
  Arms: Test implant loaded at 3 weeks post-surgery; Test implant loaded at 6 weeks post-surgery
Procedure: Early loading — Loading the implant at 3 weeks after implantation (instead of 6 weeks after implantation)
  Arms: Test implant loaded at 3 weeks post-surgery

SUMMARY:
A single centre, open, comparative, parallel group, prospective clinical investigation with a single 10 year follow up visit.

DETAILED DESCRIPTION:
This study is a continuation of two previous conducted trials:

1. Stability, long term survival and tolerability of a novel Baha® implant system, a multi-centre investigation new BIA300 (test) implant vs previous generation (control) implant:

   1. CAG5173: 6-month(1) and 3-year(2) data.
   2. CBAS5562: 5-year data(3).
2. 3 weeks loading: stability, long term survival and tolerability of a novel Baha® implant system, a multi-centre investigation 3 week loading vs 6+ week loading (= same group as control group trial 1). 6- month(4) and 3-year(5) data.

In this study the (5-year data for trial 2 and) 10-year data regarding stability, survival and soft tissue tolerability from the above mentioned trials will be evaluated and compared. The previous trials were multicentre, but the current study will be single-centred and therefore only include the participants of the Radboud site. Data will be collected at a visit at (5 years, for trial 2 and) 10 years (+/- 6 months) after implantation.

Up to now, no RCT of these implants (with the loading of 3 weeks after implantation) has assessed stability, survival and tolerability over a 10-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the original trials, patients had to be at least 18 years old.

Exclusion Criteria:

* Exclusion criteria were an inability to follow investigational procedures, any factor at the discretion of the investigator that was considered to contraindicate participation, and any disease or treatment known to compromise the bone quality at the implant site. For patients who had lost or removed the implant, the time to implant loss was recorded. Patients who could not attend the 5 or 10 year follow-up visit for other reasons were included in the implant survival analysis as well; the last available information regarding implant survival was obtained verbally from the patient, from medical records, or from information captured from the original investigations. Furthermore, patients were excluded if they had a bone thickness less than 4 mm at the implant site during implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
implant stability | 10 years after implantation
  Implant Stability Quotiënt (ISQ) will be measured at the 10y-visit. The resonance frequency analysis renders an ISQ value ranging from 1 to 100. Measurements shall be performed at the abutment level, as is done in the previous investigations. The highest and lowest ISQ value out of two perpendicular measurements shall be recorded as ISQ High and ISQ low. The measurement should preferably be done by the same Osstell instrument (Osstell, Gothenburg, Sweden) that was used in the previous completed study. SmartPeg Type 43 and 55 shall be used during the measurement (Osstell, Gothenburg, Sweden). The procedures for obtaining ISQ values is described in the manufacturer's instruction that will be handed out to the investigators.

SECONDARY OUTCOMES:
implant survival | 10 years after implantation
  All patients will be asked if they have experienced any implant osseointegration problems. The time from implantation until implant loss or removal will be noted. In case of implant removal, reason for removal shall be recorded.
soft tissue reaction | 10 years after implantation
  Soft tissue reactions will be measured using the Holgers' classification & IPS-score.
  The Holgers' classification is designed to capture signs and symptoms of inflammation or infection at the site of implantation (scale 0-4).
  The IPS-score is a complete standardized assessment scale for skin complications for both percutaneous and transcutaneous implants for bone conduction devices (BCDs) with a proposed treatment advice based on the outcome. The IPS score has three subscales: inflammation (0-4); pain (0-2), and skin height (0-2).
device use | 10 years after surgery
  To evaluate the long-term device use of a Baha®.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teunissen EM, Caspers CJI, Vijverberg MA, Mylanus EAM, Hol MKS. Long-Term Follow-up of a Wide-Diameter Bone-Anchored Hearing Implant: 10-Year Experience on Stability, Survival, and Tolerability of an Implant-Abutment Combination. Otol Neurotol. 2023 Jan 1;44(1):40-46. doi: 10.1097/MAO.0000000000003763. Epub 2022 Nov 23. PMID 36417764